CLINICAL TRIAL: NCT02704403
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of Elafibranor in Patients With Nonalcoholic Steatohepatitis (NASH) and Fibrosis
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of Elafibranor Versus Placebo in Patients With Nonalcoholic Steatohepatitis (NASH)
Acronym: RESOLVE-IT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study did not meet the predefined primary surrogate efficacy endpoint, no safety issues identified
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505-315-1; 2015-005385-38 (EudraCT Number)
Record Dates: First submitted 2016-02-16; First posted 2016-03-10 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Nonalcoholic Steatohepatitis (NASH) With Fibrosis
Keywords: Elafibranor; NASH; Nonalcoholic steatohepatitis; Fatty liver disease; Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- 120 mg Elafibranor (Experimental): Coated tablets dosed at 120mg Elafibranor; oral administration; one tablet per day before breakfast with a glass of water
  Interventions: Drug: Elafibranor
- Placebo (Placebo Comparator): Coated placebo tablets; oral administration; one tablet per day before breakfast with a glass of water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elafibranor
  Other Names: GFT505
  Arms: 120 mg Elafibranor
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the effect of Elafibranor treatment compared to placebo on 1) histological improvement and 2) all-cause mortality and liver-related outcomes in patients with nonalcoholic steatohepatitis (NASH) and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged from 18 to 75 years inclusive at first screening visit.
2. Must provide signed written informed consent and agree to comply with the study protocol.
3. Females participating in this study must be of nonchildbearing potential or using highly efficient contraception for the full duration of the study and for 1 month after the end of treatment, as described below:

   1. Cessation of menses for at least 12 months due to ovarian failure,
   2. Surgical sterilization such as bilateral oopherectomy, hysterectomy, or medically documented ovarian failure
   3. If requested by local IRB regulations and/or National laws, sexual abstinence may be considered adequate (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
   4. Using a highly effective nonhormonal method of contraception (bilateral tubal occlusion, vasectomized partner, or intra-uterine device)
   5. Double contraception with barrier AND highly effective hormonal method of contraception (oral, intravaginal, or transdermal combined estrogen and progestogen hormonal contraception associated with inhibition of ovulation; oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation; or intrauterine hormone-releasing system). The hormonal contraception must be started at least 1 month prior to Randomization.
4. Histological confirmation of steatohepatitis on a diagnostic liver biopsy by central reading of the slides (biopsy obtained within 6 months prior to randomization or during the screening period) with at least 1 in each component of the NAS score (steatosis scored 0-3, ballooning degeneration scored 0-2, and lobular inflammation scored 0-3).
5. NAS score ≥4.
6. Fibrosis stage of 1 or greater and below 4, according to the NASH CRN fibrosis staging system.
7. Stable dose of vitamin E, polyunsaturated fatty acids, or ursodeoxycholic acid from at least 6 months prior to diagnostic liver biopsy
8. For participants with type 2 diabetes, glycemia must be controlled. If glycemia is controlled by antidiabetic drugs, change in anti-diabetic therapy must follow these requirements:

   1. No qualitative change 6 months prior to diagnostic liver biopsy up to Randomization (i.e., implementation of a new anti-diabetic therapy) for participants treated with metformin, gliptins, sulfonylureas, sodium/glucose cotransporter (SGLT) 2 inhibitors, glucagon-like peptide (GLP)-1 agonists, or insulin. Dose changes of these medications are allowed in the 6 months prior to diagnostic liver biopsy, except for GLP-1 agonists, which must remain on stable dose in the 6 months prior to diagnostic liver biopsy.
   2. No implementation of GLP-1 agonists and SGLT2 inhibitors up to 72 weeks of treatment (Visit 7).

Initiation of any other antidiabetic drugs is allowed after Randomization based on treating physicians' judgment, except for glitazones which are prohibited 6 months prior to diagnostic liver biopsy until the end of treatment.

Exclusion Criteria:

1. Known heart failure (Grade I to IV of New York Heart Association classification).
2. History of efficient bariatric surgery within 5 years prior to screening.
3. Uncontrolled hypertension during the Screening Period despite optimal antihypertensive therapy
4. Type 1 diabetes participants .
5. Participants with decompensated diabetes (HbA1c>9%).
6. Participants with a history of clinically significant acute cardiac event within 6 months prior to screening
7. Weight loss of more than 5% within 6 months prior to randomization
8. Compensated and decompensated cirrhosis
9. Current or recent history (<5 years) of significant alcohol consumption
10. Pregnant or lactating females or females planning to become pregnant during the study period.
11. Other well documented causes of chronic liver disease according to standard diagnostic procedures
12. Participants with previous exposure to Elafibranor
13. Prohibited concomitant medication
14. Any medical conditions that may diminish life expectancy to less than 2 years including known cancers.
15. Evidence of any other unstable or untreated clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, neoplastic or psychiatric disease.
16. Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
17. Participants with biological criteria exclusion as per effective protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2157 (Actual)
Dates: Start 2016-03; Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Addy, MD MMSc, Study Director — Genfit
Locations (324):
- United States (152):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - The Institute for Liver Health, Chandler, Arizona
  - The Institute for Liver Health, Glendale, Arizona
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Dignity Health St. Joseph's Hospital, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Institute for Liver Health, Tucson, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - The University of Arizona College of Medicine Liver Research Institute, Tucson, Arizona
  - Liver Wellness Center, Little Rock, Arkansas
  - GW Research, Inc., Chula Vista, California
  - Southern California Research Center, Coronado, California
  - University of California, San Francisco, Fresno Community Regional Medical Center, Fresno, California
  - Fresno Clinical Research Center, Fresno, California
  - Scripps Clinic Torrey Pines, La Jolla, California
  - University of California - San Diego, La Jolla, California
  - Loma Linda University Medical Center - Transplantation Insitute, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Keck Hospital of USC, Los Angeles, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials LLC, Los Angeles, California
  - Veterans Affaires Greater Los Angeles Healthcare System, West LA VA Medical Center, Los Angeles, California
  - Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - Alliance Clinical Research, Oceanside, California
  - National Research Institute, Panorama City, California
  - Alliance Clinical Research, Poway, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of California, San Diego Airway Research and Clinical Trials Center, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - VA San Diego HealthCare System, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Sutter West Bay Hospitals dba California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, Medical Center at Parnassus, San Francisco, California
  - Ventura Clinical Trials, Ventura, California
  - South Denver Gastroenterology, Englewood, Colorado
  - Yale University School of Medicine, Section of Digestive Diseases, New Haven, Connecticut
  - Georgetown University Hospitals, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Integrity Clinical Research LLC, Doral, Florida
  - University of Florida, Gainesville, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Florida Digestive Health Specialists, LLP, Lakewood Rch, Florida
  - Atlantic Gastroenterology Associates, LLC, Lakewood Rch, Florida
  - Miami VA Healthcare System, Miami, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - University of Miami - Schiff Center for Liver Diseases, Miami, Florida
  - South Florida Center of Gastroenterology, PA, Wellington, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Summit Clinical Research, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Atlanta Medical Center, Inc., Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital - Arkes Family Pavilion, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville Medical / Dental Complex, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Kaiser Permanente Shady Grove Medical Center, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Division of Gastroenterology & Hepatology, Detroit, Michigan
  - Gastrointestinal Associates & Endoscopy Center, Flowood, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Luke's Liver Transplant & Specialist, Kansas City, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Rutgers, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Rutgers, New Jersey Medical School, Newark, New Jersey
  - Southwest Gastroenterology Associates, Albuquerque, New Mexico
  - University at Buffalo, Clinical and Translational Research Center, Buffalo, New York
  - Hofstra Northwell School of Medicine, Manhasset, New York
  - Concorde Medical Group, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York-Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - Beth Israel Medical Center, New York, New York
  - Premier Medical Group, Poughkeepsie, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - UNC Health Care System, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Gastroenterology, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Carolinas Center for Liver Disease, Carolinas HealthCare System/Atrium Health, Huntersville, North Carolina
  - Diabetes & Endocrinology Consultants, Morehead City, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Ohio Gastroenterology & Liver Institute, Cincinnati, Ohio
  - University of Cincinnati Physicians Company , LLC, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Drexel University, College of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Health System, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - UPMC Montefiore, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Associates in Gastroenterology, PLC, Hermitage, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - Baylor All Saints Medical Center - Baylor Research Institute, Fort Worth, Texas
  - DHAT Research Institute, Garland, Texas
  - Baylor College of Medicine, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - Centex Studies Inc., Houston, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - Brooke Army Medical Center, Houston, Texas
  - Gastroenterology Consultants of San Antonio, Live Oak, Texas
  - Centex Studies Inc, McAllen, Texas
  - Pinnacle Clinical Research, PLLC, Rollingwood, Texas
  - The Texas Liver Institute, Inc., San Antonio, Texas
  - Pinnacle Clinical Research, PLLC, San Antonio, Texas
  - Texas Digestive Consultants (TDDC), Southlake, Texas
  - Victoria Gastroenterology, Victoria, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Medical Campus - Center for Liver Disease, Falls Church, Virginia
  - Bon Secours Liver Institute of Virginia - Newport News, Newport News, Virginia
  - Bon Secours Liver Institute of Virginia - Richmond, Richmond, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Kaiser Permanente Springfield Medical Center, Springfield, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
- Argentina (14):
  - Sanatorio Güemes, Caba, Buenos Aires
  - Axismed S.R.L, CABA, Buenos Aires
  - Instituto de Investigaciones Clinicas San Nicolas SRL, San Nicolás de los Arroyos, Buenos Aires
  - Hospital Alemán, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular SA (CIPREC), Buenos Aires
  - Fundación Sanatorio Güemes, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Británico de Buenos Aires, Buenos Aires
  - CCBR Clinical Research, Buenos Aires
  - Centro De Hepatologia Ciudad de La Plata, La Plata
  - Hospital Universitario Austral, Pilar
  - Dim Clinica Privada, Ramos Mejía
  - Hospital Provincial del Centenario, Rosario
  - Instituto Medico Alas, Salta
- Australia (12):
  - Flinders Medical Centre, Bedford Park
  - Box Hill Hospital, Box Hill
  - Monash Medical Centre Clayton, Clayton
  - Concord Repatriation General Hospital, Concord
  - St. Vincent's Hospital Melbourne, Fitzroy
  - Austin Hospital, Heidelberg
  - Nepean Hospital, Kingswood
  - The St George Hospital, Kogarah
  - The Alfred Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Sir Charles Gairdner Hospital (SCGH), Nedlands
  - Westmead Hospital, Westmead
- Belgium (7):
  - Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier de Wallonie Picardie (CHWAPI), Tournai
- Canada (11):
  - LAIR Centre, Vancouver, British Columbia
  - Vancouver General Hospital (VGH) - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Monteregie Centre de Recherche, Greenfield Park, Quebec
  - The Montreal Chest Institute, Montreal, Quebec
  - University of Calgary, Cumming School of Medicine, Calgary, AB
  - Queen Elizabeth II Health Sciences Centre, Nova Scotia Health Authority, Halifax
  - Mc Gill University Health Centre (MUHC), Montreal
  - University of Manitoba, Winnipeg, MB
- Chile (6):
  - Hospital de La Serena, La Serena
  - Alta Salud, Los Ángeles
  - Hospital Clínico UC, Santiago
  - Hospital Clínico Universidad de Chile, Santiago
  - Centro de Estudios Clinicos Barros Luco SPA (Patients seen, Fibroscan stored and Drug Shipment), Santiago
  - Clínica Reñaca, Viña del Mar
- Colombia (7):
  - Solano&Terront Servicios Médicos LTDA - Unidad Integral de Endocrinologia UNIENDO, Bogotá, Bogota D.C.
  - Fundación Cardio Infantil - Instituto de Cardiología, Bogotá
  - Fundación Valle del Lili, Cali
  - Centro Medico Imbanaco, Cali
  - Fundacion Hospitalaria San Vicente de Paul, Medellín
  - Hospital Universitario San Vicente de Paul Fundación, Medellín
  - Hospital Pablo Tobon Uribe, Medellín
- Czechia (4):
  - Fakultní Nemocnice Brno, Brno
  - Research Site S.R.O., Pilsen
  - Research Site, s.r.o, Pilsen
  - KlinMed s.r.o., Prague
- Aarhus University Hospital, Aarhus, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- France (18):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - Hôpital Antoine-Béclère, Clamart
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Saint Joseph, Marseille
  - CHRU Montpellier- Hôpital Saint Eloi, Montpellier
  - CHU de Nantes - Hôpital Laennec, Nantes
  - CHU de Nice- Hôpital de l'Archet II, Nice
  - Hôpital Saint-Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hôpital Cochin, Paris
  - Hôpital Haut-Lévêque, Pessac
  - CHU Toulouse - Hôpital Purpan, Toulouse
  - CHU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse, Villejuif
- Germany (18):
  - Universitätsklinikum Köln, Cologne, Northwest
  - Universitätsklinikum RWTH Aachen, Aachen
  - Liver Center, Berlin
  - Gastroenterologie am Bayerischen Platz/ Gastro-Studien, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt - Goethe Universität, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - EUGASTRO GmbH, Leipzig
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Würzburg, Würzburg
- Italy (8):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Policlinico Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Casa Sollievo della Sofferenza I.R.C.C.S., San Giovanni Rotondo
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino - Ospedale Molinette, Torino
- Mexico (6):
  - Hospital Angeles Clinica Londres, México, DIF
  - Centro de Investigación Clínica del Pacífico, S.A de C.V., Acapulco
  - Hospital Maria Auxiliadora, Guadalajara
  - Médica Sur, Mexico City
  - Consultorio Medico, Mexico City
  - Accelerium S de RL de C.V., Monterrey
- Netherlands (4):
  - Vrije Universiteit Medical Center, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Maastricht UMC+, Maastricht
  - Radboud UMC, Nijmegen
- Portugal (6):
  - Centro Hospitalar e Universitário de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar Lisboa Central, EPE - Hospital Santo António dos Capuchos, Lisbon
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital Santa Maria, Lisbon
  - Centro Hospitalar de São João, EPE - Hospital de São João, Porto
  - Centro Hospitalar de São João, Porto
  - Centro Hospita de Tras-os-Montes e Alto Douro, EPE, Vila Real
- Puerto Rico (4):
  - Caparra Internal Medicine Research Center, Río Grande
  - Klinical Investigations Group, LLC, San Juan
  - Fundacion de Investigacion de Diego, San Juan
  - Fundación de Investigación, San Juan
- Romania (4):
  - Institutul National de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - SC Cabinet Particular Policlinic Algomed SRL, Timișoara
  - Spitalul Clinic Judetean de Urgenta "Pius Brinzeu" Timisoara, Timișoara
- Russia (6):
  - FSBRI "Federal Research Center of nutrition and biotechnology, Moscow
  - I. M. Sechenov - First Moscow State Medical University, Moscow
  - M. F. Vladimirsky - Clinical Research Institution of Moscow Region, Moscow
  - Military medical academy n. a. S.M. Kirov, Saint Petersburg
  - City Clinical Hospital No. 31, Saint Petersburg
  - St Petersburg State Budgetary Healthcare Institution City Clinical Hospital N°31, Saint Petersburg
- South Africa (3):
  - Tiervlei Trial Centre, Cape Town
  - Mediclinic Constantiaberg, Cape Town
  - Phoenix Pharma (Pty) Ltd, Port Elizabeth
- Spain (9):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Campus Hospital Universitario Virgen del Rocío - Instituto de Biomedicina de Sevilla (IBIS), Seville
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden
- Switzerland (4):
  - INSELSPITAL, University Hospital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich
- Turkey (Türkiye) (6):
  - Ankara Üniversitesi Tıp Fakültesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi, Çapa
  - Bezmiâlem Vakıf Üniversitesi, Fatih
  - Sağlık Bilimleri Üniversitesi Ümraniye Eğitim ve Araştırma Hastanesi, Istanbul
  - Ege Üniversitesi, Izmir
  - Marmara Üniversitesi Eğitim ve Araştırma Hastanesi, Pendik
- United Kingdom (12):
  - University Hospitals Birmingham NHS foundation Trust, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Frimley Park Hospital NHS Foundation Trust, Frimley
  - Hull and East Yorkshire Hospitals NHS Trust - Hull Royal Infirmary, Hull
  - Bart Health NHS Trust- Royal London Hospital, London
  - The Royal Free London NHS Foundation Trust - The Royal Free Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust - St Thomas' Hospital, London
  - St George's University Hospitals NHS Foundation Trust - St George's Hospital, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS FoundationTrust - Queen's Medical Centre, Nottingham
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth
  - Portsmouth Hospitals NHS Trust - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The version 3 protocol for Brazil is included in the uploaded documents as it was part of the pre-specified plan, but this country was not used as part of the study.
Groups:
- 120 mg Elafibranor: Coated 120mg elafibranor tablets; oral administration; one tablet per day before breakfast with a glass of water
Period: Overall Study
Arm/Group | 120 mg Elafibranor | Placebo
Started | 1437 | 720
Full Intent-to-Treat Population | 1437 | 720
Full Safety Population | 1433 | 717
Completed | 0 | 0
Not Completed | 1437 | 720
Not completed — Randomized and not treated (due to non-compliance with protocol) | 4 | 3
Not completed — Administrative reasons by sponsor | 1251 | 616
Not completed — Death | 4 | 3
Not completed — Endpoint event | 52 | 24
Not completed — Lost to Follow-up | 22 | 11
Not completed — Protocol Violation | 15 | 15
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 85 | 45
Not completed — Investigator decision | 1 | 1
Not completed — Follow-up not possible | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 120 mg Elafibranor | Placebo | Total
Number analyzed (Participants) | 1437 | 720 | 2157
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.78) | 54.4 (11.63) | 54.1 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 622 | 308 | 930
  Male | 815 | 412 | 1227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 336 | 177 | 513
  Not Hispanic or Latino | 1089 | 532 | 1621
  Unknown or Not Reported | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 1 | 9
  Asian | 53 | 27 | 80
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 28 | 10 | 38
  White | 1234 | 614 | 1848
  More than one race | 93 | 49 | 142
  Unknown or Not Reported | 18 | 16 | 34
Weight [Mean (Standard Deviation); unit: kg] | 98.0 (21.90) | 96.3 (20.84) | 97.4 (21.56)
Height [Mean (Standard Deviation); unit: cm] — Population: All participants with data available are presented
  cm
    number analyzed (Participants) | 1436 | 718 | 2154
    (all) | 169.1 (10.48) | 168.8 (10.23) | 169.0 (10.39)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: All participants with data available are presented
  kg/m^2
    number analyzed (Participants) | 1436 | 718 | 2154
    (all) | 34.1 (6.13) | 33.6 (5.77) | 33.9 (6.01)
Waist Circumference [Mean (Standard Deviation); unit: cm] — Population: All participants with data available are presented
  cm
    number analyzed (Participants) | 1431 | 719 | 2150
    (all) | 111.9 (14.19) | 110.4 (13.48) | 111.4 (13.97)
Child Bearing Potential [Count of Participants; unit: Participants]
  Yes | 105 | 46 | 151
  No | 516 | 262 | 778
  Not applicable | 815 | 412 | 1227
  Missing | 1 | 0 | 1
Type 2 Diabetes [Count of Participants; unit: Participants]
  Yes | 699 | 351 | 1050
  No | 738 | 369 | 1107
Fibrosis Stage [Count of Participants; unit: Participants] — There are five stages of fibrosis with F0: no scarring (no fibrosis); F1: minimal scarring; F2: scarring has occurred and extends outside the liver area (significant fibrosis); F3: fibrosis spreading and forming bridges with other fibrotic liver areas (severe fibrosis); F4: cirrhosis or advanced scarring.
  Participants
    F1 | 135 | 69 | 204
    F2 | 603 | 302 | 905
    F3 | 699 | 349 | 1048
Non-alcoholic fatty liver disease Activity Score Grouped Severity Score (categorical) [Count of Participants; unit: Participants] — Non-alcoholic fatty liver disease Activity Score Severity Score (NAS score) is a measure of grade and is the sum of numerical scores applied to steatosis (0-3), hepatocellular ballooning (0-2), and lobular inflammation (0-3). Accordingly, the NAS ranges from 0 to 8.
  NAS scores of 0-2 are considered not diagnostic of NASH, NAS scores of 3-4 are considered as NASH diagnostic, borderline, or positive for NASH.
  NAS Scores of 5-8 occurred in cases that are largely considered diagnostic of NASH
  Participants
    Moderate (4-5) | 663 | 317 | 980
    Severe (greater than or equal to 6) | 774 | 402 | 1176
Non-alcoholic fatty liver disease Activity Score Severity Score (categorical) [Count of Participants; unit: Participants] — Non-alcoholic fatty liver disease Activity Score Severity Score (NAS score) is a measure of grade and is the sum of numerical scores applied to steatosis (0-3), hepatocellular ballooning (0-2), and lobular inflammation (0-3). Accordingly, the NAS ranges from 0 to 8.
  NAS scores of 0-2 are considered not diagnostic of NASH, NAS scores of 3-4 are considered as NASH diagnostic, borderline, or positive for NASH.
  NAS Scores of 5-8 occurred in cases that are largely considered diagnostic of NASH
  Participants
    4 | 193 | 94 | 287
    5 | 470 | 223 | 693
    6 | 453 | 225 | 678
    7 | 271 | 154 | 425
    8 | 50 | 23 | 73
    Missing | 0 | 1 | 1
Model For End-Stage Liver Disease Score (categorical) [Count of Participants; unit: Participants] — The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease. the score is useful both in predicting short-term survival in groups of patients on the waiting list for liver transplantation as well as the risk of postoperative mortality. Patients are assigned a score from 6 to 40, with 40 representing the greatest severity of liver disease, and a high risk of death in the ensuing three months without transplantation. Patients with score < 15 are deferred of liver transplantation.
  Participants
    Less than 15 | 1426 | 715 | 2141
    Greater than or equal to 15 | 11 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Elafibranor-treated Participants Relative to Placebo Achieving Resolution of Nonalcoholic Steatohepatitis Without Worsening of Fibrosis
Description: To evaluate the effect of Elafibranor compared to placebo on liver histology in nonalcoholic steatohepatitis (NASH) participants with fibrosis by assessing the following endpoint: The number of Elafibranor-treated participants relative to placebo achieving NASH resolution without worsening of fibrosis. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurement at 72 weeks
Population: Intent-to-treat Set: a cohort of randomized F2 to F3 participants who completed the Week 72 treatment period or discontinued the study treatment early.
Measure: Count of Participants; unit: Participants
Groups:
- 120 mg Elafibranor: Coated 120 mg elafibranor tablets; oral administration; one tablet per day before breakfast with a glass of water
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 717 | 353
Participants | 138 | 52
Statistical Analysis 1: Comparison: 120 mg Elafibranor vs Placebo; The null hypothesis was that there was no difference in response rates between the elafibranor and placebo treatment groups. The alternative hypothesis was that there was a difference in the response rates between the elafibranor and placebo treatment groups; Test type: Superiority; p = 0.0659, Regression, Logistic; test is 2-sided, alpha=0.01; Mean Difference (Net) = 0.043, 95% CI 2-sided [-0.003 to 0.090]

2. Primary Outcome: Time to Long-term Outcome Composed of All-cause Mortality, Cirrhosis, and Liver-related Clinical Outcomes
Description: Composite long-term outcome measured by the number of participants with the onset of any of the adjudicated events, composed of death due to any cause, histological liver cirrhosis, and the full list of portal hypertension/cirrhosis related events as follows: liver transplantation; model for end stage liver disease (MELD) score greater than or equal to 15 for participants with baseline score less than or equal to 12, and onset of variceal bleeding requiring hospitalization, hepatic encephalopathy with West Haven/Conn score greater than or equal to 2 and requiring hospitalization, spontaneous bacterial peritonitis, and ascites requiring treatment. The MELD scale ranges from 6 to 40, showing how much a participant needs a liver transplant: higher number is more urgent. The West Haven/Conn scale is 5-point (0 to 4) grading severity of hepatic encephalopathy: higher score means worse hepatic encephalopathy. This outcome measure is for the long-term endpoint analysis.
Time Frame: From first randomization up to early termination of the study corresponding to 54 months (54 months being the longest duration for any given participant)
Population: Full Intent-to-Treat Set: All randomized participants. Participants were analyzed according to their randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 1437 | 720
Participants
  Baseline: Events | 0 | 0
  Baseline: Censored | 0 | 0
  Baseline: No events or not censored | 1437 | 720
  6 months: Events | 1 | 1
  6 months: Censored | 48 | 26
  6 months: No events or not censored | 1388 | 693
  12 months: Events | 1 | 1
  12 months: Censored | 159 | 82
  12 months: No events or not censored | 1277 | 637
  18 months: Events | 53 | 28
  18 months: Censored | 374 | 195
  18 months: No events or not censored | 1010 | 497
  24 months: Events | 56 | 31
  24 months: Censored | 609 | 301
  24 months: No events or not censored | 772 | 388
  30 months: Events | 57 | 31
  30 months: Censored | 778 | 393
  30 months: No events or not censored | 602 | 296
  36 months: Events | 60 | 32
  36 months: Censored | 1049 | 531
  36 months: No events or not censored | 328 | 157
  42 months: Events | 61 | 32
  42 months: Censored | 1293 | 652
  42 months: No events or not censored | 83 | 36
  48 months: Events | 61 | 32
  48 months: Censored | 1374 | 687
  48 months: No events or not censored | 2 | 1
  54 months: Events | 61 | 32
  54 months: Censored | 1376 | 688
  54 months: No events or not censored | 0 | 0
Statistical Analysis 1: Comparison: 120 mg Elafibranor vs Placebo; Test type: Superiority; Cox Proportional Hazard = 0.950, 95% CI 2-sided [0.619 to 1.457] — No formal test due to the early termination of the study

3. Secondary Outcome: Number of Elafibranor-treated Participants Relative to Placebo Achieving Improvement of Fibrosis of at Least 1 Stage
Description: To evaluate the effect of Elafibranor compared to placebo on liver histology in nonalcoholic steatohepatitis (NASH) participants by assessing the following endpoint: The number of Elafibranor-treated participants relative to placebo achieving improvement of liver fibrosis of at least 1 stage according to NASH Clinical Research Network (CRN) Scoring. As the primary efficacy objective was not met, the secondary efficacy endpoints were not formally tested. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurements at 72 weeks
Population: Intent-to-Treat Set: For the purpose of analysis sets aligned with efficacy summaries, a cohort of randomized F2 to F3 participants who completed the Week 72 treatment period or discontinued the study treatment early were considered.
Measure: Count of Participants; unit: Participants
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 717 | 353
Participants | 176 | 79

4. Secondary Outcome: Change From Baseline of Hemoglobin A1c (HbA1c) in Diabetic Participants After 72 Weeks of Treatment in Elafibranor-treated Participants Relative to Placebo
Description: Hemoglobin A1c (HbA1c) were tested at Week 72. Changes from baseline in HbA1c at Week 72 were evaluated. As the primary efficacy objective was not met, the secondary efficacy endpoints were not formally tested. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurements after 72 weeks of treatment and up to study termination
Population: Intent-to-Treat Set: a cohort of randomized F2 to F3 participants who completed the Week 72 treatment period or discontinued the study treatment early. Number of participants with diabetes who had available data at Week 72 are presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 318 | 150
mmol/L | 0.03 [-0.19 to 0.25] | -0.01 [-0.24 to 0.23]

5. Secondary Outcome: Change From Baseline of High-density Lipoprotein (HDL) Cholesterol After 72 Weeks of Treatment in Elafibranor-treated Participants Relative to Placebo
Description: High-density lipoprotein (HDL) cholesterol was tested at Week 72. Changes from baseline in HDL cholesterol were evaluated at Week 72. As the primary efficacy objective was not met, the secondary efficacy endpoints were not formally tested. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurements after 72 weeks of treatment and up to study termination
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 629 | 303
mmol/L | -0.036 [-0.050 to -0.021] | -0.052 [-0.073 to -0.032]

6. Secondary Outcome: Change From Baseline of Low-density Lipoprotein (LDL) Cholesterol After 72 Weeks of Treatment in Elafibranor-treated Participants Relative to Placebo
Description: Low-density lipoprotein (LDL) cholesterol was tested at Week 72. Changes from baseline in LDL cholesterol were evaluated at Week 72. As the primary efficacy objective was not met, the secondary efficacy endpoints were not formally tested. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurements after 72 weeks of treatment and up to study termination
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 600 | 283
mmol/L | -0.250 [-0.295 to -0.204] | -0.217 [-0.282 to -0.151]

7. Secondary Outcome: Change From Baseline of Homeostatic Model Assessment-IR (HOMA-IR) After 72 Weeks of Treatment in Elafibranor-treated Participants Relative to Placebo in Non-diabetic Participants
Description: Homeostatic model assessment-IR (HOMA-IR) was tested at Week 72. Changes from baseline in HOMA-IR were evaluated at Week 72. As the primary efficacy objective was not met, the secondary efficacy endpoints were not formally tested. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurements after 72 weeks of treatment and up to study termination
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 311 | 152
index | -0.789 [-2.979 to 1.402] | -0.930 [-3.347 to 1.486]

8. Secondary Outcome: Change From Baseline of Non-high Density Lipoprotein Cholesterol After 72 Weeks of Treatment in Elafibranor-treated Participants Relative to Placebo
Description: Non-high density lipoprotein (HDL) cholesterol was tested at Week 72. Changes from baseline in non-HDL cholesterol were evaluated at Week 72. As the primary efficacy objective was not met, the secondary efficacy endpoints were not formally tested. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurements after 72 weeks of treatment and up to study termination
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 609 | 302
mmol/L | -0.445 [-0.499 to -0.392] | -0.271 [-0.348 to -0.195]

9. Secondary Outcome: Change From Baseline of Triglycerides After 72 Weeks of Treatment in Elafibranor-treated Participants Relative to Placebo
Description: Triglycerides was tested at Week 72. Changes from baseline in triglycerides were evaluated at Week 72. As the primary efficacy objective was not met, the secondary efficacy endpoints were not formally tested. This outcome measure is for the surrogate endpoint analysis.
Time Frame: Measurements after 72 weeks of treatment and up to study termination
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 120 mg Elafibranor | Placebo
Number analyzed (Participants) | 636 | 307
mmol/L | -0.466 [-0.537 to -0.395] | -0.148 [-0.249 to -0.046]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected at every study visit from screening up to early termination of the study corresponding to 54 months (54 months being the longest duration for any given participant) plus 30 days.
Description: The 9 deaths reported in the all cause mortality section correspond to all death events adjudicated throughout the study duration. Among the 9 deaths, 7 deaths (4 in elafibranor arm; 3 in the placebo arm) resulted in early study discontinuation of participants in the Full Safety Population, as reported in the Participant Flow section.
Arm/Group | 120 mg Elafibranor | Placebo
All-Cause Mortality (participants affected / at risk) | 6/1437 | 3/720
Serious Adverse Events (participants affected / at risk) | 190/1433 | 95/717
Other Adverse Events (participants affected / at risk) | 1227/1433 | 601/717
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 120 mg Elafibranor (N=1433) | Placebo (N=717)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 5 (6)
Acute myocardial infarction (Cardiac disorders) | 5 | 0
Cardiac failure (Cardiac disorders) | 2 (4) | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac asthma (Cardiac disorders) | 1 (3) | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 (2)
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 1 | 0
Primary hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Pancreatitis acute (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Ileus (Gastrointestinal disorders) | 2 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 1 | 0
Coeliac artery stenosis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 5 | 2
Chest pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Gallbladder necrosis (Hepatobiliary disorders) | 0 | 1
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 3 (5)
Diverticulitis (Infections and infestations) | 5 | 2
Cellulitis (Infections and infestations) | 3 | 2 (3)
Urinary tract infection (Infections and infestations) | 2 | 3
Appendicitis (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 (2) | 0
Abscess limb (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 1 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 1
Infected bite (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Shigella sepsis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Bladder injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Chest crushing (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 (6)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (5) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian endometrioid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 4 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Lumbar radiculopathy (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 2 | 0
Meningocele acquired (Nervous system disorders) | 1 (2) | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Vertebral artery dissection (Nervous system disorders) | 0 | 1
Wernicke-Korsakoff syndrome (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device malfunction (Product Issues) | 1 (3) | 0
Device loosening (Product Issues) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 (2) | 1
Major depression (Psychiatric disorders) | 1 (2) | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Renal colic (Renal and urinary disorders) | 3 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 (4) | 0
Hypertension (Vascular disorders) | 1 (3) | 0
Aortic dissection (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 120 mg Elafibranor (N=1433) | Placebo (N=717)
Diarrhoea (Gastrointestinal disorders) | 148 (171) | 68 (82)
Nausea (Gastrointestinal disorders) | 140 (158) | 50 (51)
Abdominal pain upper (Gastrointestinal disorders) | 83 (105) | 47 (49)
Abdominal pain (Gastrointestinal disorders) | 79 (94) | 49 (57)
Fatigue (General disorders) | 103 (111) | 49 (54)
Urinary tract infection (Infections and infestations) | 145 (236) | 77 (134)
Nasopharyngitis (Infections and infestations) | 134 (186) | 52 (61)
Influenza (Infections and infestations) | 115 (127) | 54 (68)
Upper respiratory tract infection (Infections and infestations) | 107 (132) | 46 (55)
Bronchitis (Infections and infestations) | 93 (111) | 33 (36)
Sinusitis (Infections and infestations) | 72 (96) | 43 (53)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 102 (109) | 58 (62)
Arthralgia (Musculoskeletal and connective tissue disorders) | 160 (202) | 81 (110)
Back pain (Musculoskeletal and connective tissue disorders) | 120 (144) | 60 (62)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 71 (77) | 25 (27)
Headache (Nervous system disorders) | 98 (114) | 43 (46)
Cough (Respiratory, thoracic and mediastinal disorders) | 85 (99) | 40 (47)
Hypertension (Vascular disorders) | 86 (99) | 39 (42)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated based upon limited efficacy at time of the interim analysis, not due to safety concerns, and the conclusion that there would be limited benefit for participants to continue in the trial. Therefore, the results for efficacy endpoints other than the primary and key secondary endpoints are not presented in the disclosure of these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All materials, information (oral or written) and unpublished documentation provided to the Investigators (or any company/institution acting on their behalf) are the exclusive property of the Sponsor and may not be given or disclosed, either in part or in whole, by the Investigator or by any person under his/her authority to any third party without the prior express consent of the Sponsor.

DOCUMENTS (3):
  • Study Protocol: Local Protocols (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT02704403/Prot_000.pdf
  • Study Protocol: General Protocols (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT02704403/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT02704403/SAP_002.pdf